CLINICAL TRIAL: NCT02858700
Title: Value for Cord Blood Procalcitonin to Diagnose Early Neonatal Bacterial Infection
Acronym: PCT_CORDON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8271
Record Dates: First submitted 2016-07-21; First posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Neonatal Bacterial Infection
Keywords: neonatal bacterial infection; procalcitonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- umbilical cord blood procalcitonin (Experimental): dosage of the umbilical cord blood Procalcitonin for diagnosing of IBNP
  Interventions: Biological: dosage of the umbilical cord blood Procalcitonin for diagnosing of IBNP

INTERVENTIONS:
Biological: dosage of the umbilical cord blood Procalcitonin for diagnosing of IBNP

SUMMARY:
After birth, in the presence of risk factors for early neonatal bacterial infection (IBNP), the pediatrician must make a difficult decision quickly or not to prescribe additional examinations and / or hospitalize or not the newborn in order to administer parenteral antibiotics. This decision takes into account several contextual data, (clinical, biological and bacteriological clinical data) to be considered simultaneously. These information lack sensitivity and specificity.

Therefore, the common attitude among newborns in many countries remains the achievement of a significant number of additional tests and the establishment, without a prior evidence of infection, intravenous empirical antibiotic therapy for 48 -72h at least in hospitalization. However, the diagnosis of IBNP posteriori, is often reversed. This attitude is:

1. one source to higher health care costs (hospitalization, additional examinations)
2. Selection of the bacterial ecology of the newborn and neonatal services and
3. stress for the newborn and parents

ELIGIBILITY:
Inclusion Criteria:

* Birth to motherhood.
* Term > 34 weeks .
* Presence of at least one of the factors of major or minor infection risk

Exclusion Criteria:

* cord blood sample unavailable.
* Death in the delivery room
* Corticosteroids prenatally (modification of cytokine production ) .

Ages: 1 Minute to 30 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 550 (Actual)
Dates: Start 2009-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
value of the procalcitonin in the umbilical cord blood | up to 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided